CLINICAL TRIAL: NCT03609281
Title: Cesarean Scar Characteristics After Scheduled and Emergency Cesarean Deliveries: A Single Center Study
Brief Title: Cesarean Scar Characteristics After Scheduled and Emergency Cesarean Deliveries
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Prinicipal investigator, Tanta University
Other Study IDs: Ayman CS Scar
Record Dates: First submitted 2018-07-15; First posted 2018-08-01 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Cesarean Scar Niche; Cesarean Wound; Dehiscence; Cesarean Section; Dehiscence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scheduled cesaren group: Patient delivered by elective cesarean section without labour pains
  Interventions: Radiation: Ultrasound assessement of uterine scar
- Emergency cesarean group: Patients delivered by cesarean section due to an emergency
  Interventions: Radiation: Ultrasound assessement of uterine scar

INTERVENTIONS:
Radiation: Ultrasound assessement of uterine scar — 3D ultrasound assessment of scar characteristics

SUMMARY:
This study was designed to evaluate the scar characteristics following scheduled and emergency cesarean deliveries.

DETAILED DESCRIPTION:
design and settings: This study is a descriptive, cross-sectional and multicenter study conducted at Tanta and Benha Universities, Egypt in the period from August, 1, 2018 to December, 31, 2018.

Patients:

Eligibility: Nine hundred patients were selected carefully according to inclusion and exclusion criteria. The inclusion criteria were: (i) Primipara having prior cesarean delivery whether scheduled or emergency (ii) Term delivery ≥ 37 weeks of gestation (iii) Multipara having the last delivery by cesarean either scheduled or emergency (iv) The interval following cesarean delivery to be 6 months at least and (v) Double-layer repair of uterus and (vi) Cesarean by pfannensteil incisions. The exclusion criteria were: (i) Repeat cesarean sections (ii) Preterm delivery (iii) Associated placental abnormalities (iv) Single-layer repair of uterus and (v) Refusal to participate.

Allocations: This study is not a clinical trial so allocation is made based on characteristics of patients and eligibility to be allocated in either scheduled cesarean group or emergency cesarean group. The allocation was not equal based on the percentage of patients in either group. The scheduled cesarean group included 580 cases while the emergency cesarean group included 320 cases from both universities.

Intervention: Cesarean scar assessment included both uterine scar and cutaneous scar. The uterine scar was assessed by transvaginal 3D ultrasound. The used device in both universities was DC-30 device of Mindray Company. All ultrasound examinations were conducted by third author in this study. Cutaneous scar was assessed by surgery department represented by the fourth author in this study. The uterine scar in both groups was examined for distance from internal os, length, thickness, volume, vasculature and presence of any defects. Cutaneous scar was examined for distance from symphysis pubis, length, shape, any depressed areas, any defects (hernia orifice), sinus and presence of keloid or hypertrophic scar.

ELIGIBILITY:
Inclusion Criteria:

* Primipara delivered by cs
* Multipara with last delivery by cs
* Full term delivery >37 weeks
* Double layer cesarean repair
* Pfannenstiel incison

Exclusion Criteria:

* Repeat cs
* Any placental abnormalities
* Preterm delivery
* Single layer cesarean repair
* Refusal to participate

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients will be selected according to inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Scar characteristics | 6 months
  Site of scar in relation to internal os of cervix
Scar length | 6 months
  length of scar in mm
thickness of scar | 6 months
  Scar depth in mm
Scar volume | 6 months
  Length multiplied by width multiplied by depth
Scar vascularity | 6 month
  Doppler on scar to assess vascularity

SECONDARY OUTCOMES:
Scar defect or niche | 6 months
  Assessment of scar weakness or scar defect by ultrasound with measurement of depth, width and length of defects plus the residual myometrial tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) are secret